CLINICAL TRIAL: NCT04716712
Title: Mortalite Infantile Reduite Par l'Administration de Masse de l'Azitromycine
Brief Title: Infant Mortality Reduction by the Mass Administration of Azithromycin
Acronym: MIRAMA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Helen Keller International (Other); Centre de Recherche en Sante de Nouna, Burkina Faso (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-32979
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Child Mortality
Keywords: Azithromycin; Mass Drug Administration; Child Mortality
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: The study will be a double-blind, placebo-controlled, cluster-randomized trial in which health centers (CSPS) in the 3 intervention regions will be randomized to either CHD combined with placebo (33%) or CHD combined with Azithromycin (67%), an allocation of 1:2 that favors active treatment. The allocation sequence and treatment labels will be masked to all but one biostatistician and one analyst at UCSF. The placebo will be indistinguishable from the active azithromycin.
  Antimicrobial resistance will be monitored in a parallel study of communities from the target study area. 60 communities will be randomly selected among eligible communities, and randomized in a 1 : 1 fashion to CHD+placebo or CHD+azithromycin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a quadruple blinded study. Only one biostatistician and one analyst at UCSF will have the unmasking information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Biannual mass oral azithromycin + child health days (Active Comparator): Bi-annual Mass Azithromycin distribution to all children 1-11 months old in participating communities paired with the Child Health Days Vitamin A distribution platform
  Interventions: Drug: Azithromycin
- Biannual mass placebo + child health days (Placebo Comparator): Bi-annual Mass placebo distribution to all children 1-11 months old in participating communities paired with the Child Health Days Vitamin A distribution platform
  Interventions: Drug: Placebo
- Resistance Sub Study: Azithromycin + Child Health Days (Active Comparator): Antimicrobial resistance will be monitored in a parallel study of communities from the target study area. 60 communities will be randomly selected among eligible communities, and randomized in a 1 : 1 fashion
  Interventions: Drug: Azithromycin
- Resistance Sub Study: Placebo + Child Health Days (Placebo Comparator): Antimicrobial resistance will be monitored in a parallel study of communities from the target study area. 60 communities will be randomly selected among eligible communities, and randomized in a 1 : 1 fashion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin is a macrolide-type antibiotic that is used to treat various types of infections. Previous studies in Niger have demonstrated a nearly 18% reduction in all-cause child mortality following biannual mass administration to children 1-59 months.
  Other Names: Zithromax
  Arms: Biannual mass oral azithromycin + child health days; Resistance Sub Study: Azithromycin + Child Health Days
Drug: Placebo — Matching identical placebo in packaging, appearance, and taste.
  Arms: Biannual mass placebo + child health days; Resistance Sub Study: Placebo + Child Health Days

SUMMARY:
This trial will investigate the supplementation of azithromycin distribution to the "Child Health Days" platform in Burkina Faso for child mortality reduction. This distribution will pair door-to-door administration of vitamin A and azithromycin or placebo with acute malnutrition screening among children 1-11 months old.

DETAILED DESCRIPTION:
The MORDOR clinical trial funded by the Bill & Melinda Gates Foundation in Malawi, Tanzania, and Niger demonstrated that biannual oral azithromycin distributions to children aged 1-59 months significantly reduced child mortality. The investigators hypothesize that biannual administration of azithromycin to children aged 1-11 months will reduce mortality in this age group. The aim of the project is to demonstrate that this intervention can be scaled up and produce the same benefits on mortality as those documented in smaller, more controlled studies. Since 1986, to reduce child mortality, Burkina Faso has been administering high-dose vitamin A supplementation to children aged 6-59 months on a biannual basis through the "Child Health Days" platform. The "Child Health days" are a door-to-door distribution of vitamin A coupled with screening for acute malnutrition in children aged 6-59 months and deworming of children aged 12-59 months. This approach has been successful but expensive. A new strategy implemented since September 2017 relies on community-based health workers (CBHWs) to distribute Vitamin A in rural areas, and on community-based distributors (CDs) in urban areas. Based on expert opinion and the preliminary findings of formative research conducted by the Ministry of Health and Helen Keller International, it was agreed that the Child Health Days platform was the most appropriate platform to implement the biannual administration of azithromycin to children aged 1 to 11 months.

In this trial, mortality will be measured via complete birth history which will be collected in a subset of villages in the study area before the first treatment distribution. The study team will also conduct a baseline census of the study areas for treatment coverage estimations.

Sixty villages (30 azithromycin, 30 placebo) will contribute to the macrolide resistance outcomes, where the study team will collect rectal and nasal swabs from children 1-59 months.

ELIGIBILITY:
Inclusion Criteria:

Community eligibility criteria:

* Located in one of the three selected regions: SudOuest, Centre-Ouest, Hauts-Bassins
* Verbal consent of the community leader is obtained

Inclusion criteria for children:

* Aged 1 to 11 months
* Living in one of the communities participating in the study

Exclusion Criteria:

Community exclusion criteria:

• Inaccessible or unsafe for the study team

Exclusion criteria for children:

• Known allergy to macrolides

Ages: 1 Month to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 694400 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 24 months following baseline
  a) Evaluate whether azithromycin integrated within the VAD+ platform reduces mortality in children aged 1-11 months old compared to placebo

SECONDARY OUTCOMES:
Antimicrobial Resistance (AMR) | 24 months
  b) To compare the cluster level load of genetic determinants of macrolides resistance in rectal samples collected from children 1-59 months old in the clusters receiving azithromycin compared to the clusters receiving placebo
Clinic Visits | 24 months
  b) Evaluate whether azithromycin integrated within the VAD+ platform changes the rate of clinic visits in children aged 1-11 month old compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lietman, MD, Principal Investigator — University of California, San Francisco; Georges Dimithe, Study Director — Helen Keller International
Locations (3):
- University of California, San Francisco, San Francisco, California, United States
- Burkina Faso (2):
  - Centre de Recherche en Sante de Nouna, Nouna
  - Helen Keller International, Ouagadougou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keenan JD, Bailey RL, West SK, Arzika AM, Hart J, Weaver J, Kalua K, Mrango Z, Ray KJ, Cook C, Lebas E, O'Brien KS, Emerson PM, Porco TC, Lietman TM; MORDOR Study Group. Azithromycin to Reduce Childhood Mortality in Sub-Saharan Africa. N Engl J Med. 2018 Apr 26;378(17):1583-1592. doi: 10.1056/NEJMoa1715474. PMID 29694816
- [Derived] Yago-Wienne F, Toure D, Dimithe G, Khassanova R, Sidibe S, Some PN, Bamba I, Zombre V, Sie A, Bountogo M, Coulibaly B, Ouattara M, Peterson B, Arnold B, Lietman TM, Lebas E, O'Brien KS. Integration of azithromycin mass administration to 1-11-month-old children into an existing health platform to reduce child mortality: a cluster-randomised trial in Burkina Faso. BMJ Glob Health. 2026 Jan 8;11(1):e021336. doi: 10.1136/bmjgh-2025-021336. PMID 41506755